CLINICAL TRIAL: NCT01404507
Title: Efficacy of Combination of IntraCoronary Bolus Abciximab and Aspiration Thrombectomy in Patients With Acute ST-segment Elevation Myocardial Infarction; ICAT Trial
Brief Title: Efficacy of Combination of IntraCoronary Bolus Abciximab and Aspiration Thrombectomy in STEMI
Acronym: ICAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Korean Society of Interventional Cardiology (Unknown)
Responsible Party: Principal Investigator, Sung Gyun Ahn, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICAT_ver_1.2
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction
MeSH Terms: interventions — Abciximab; Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intracoronary abciximab (Active Comparator): Intracoronary injection of bolus abciximab
  Interventions: Drug: Gp 2b 3a inhibitor
- Aspiration thrombectomy (Active Comparator): Aspiration thrombectomy
  Interventions: Device: aspiration thrombectomy
- Both use (Active Comparator): Both use of intracoronary injection of bolus abciximab and aspiration thrombectomy
  Interventions: Other: Both use

INTERVENTIONS:
Drug: Gp 2b 3a inhibitor — bolus injection of abciximab via intracoronary route single injection during primary PCI dosage : 0.25mg/kg
  Other Names: clotinab
  Arms: Intracoronary abciximab
Device: aspiration thrombectomy — Aspiration thrombectomy via aspiration catheter
  Other Names: Thrombuster II
  Arms: Aspiration thrombectomy
Other: Both use — Both use of intracoronary abciximab and aspiration thrombectomy
  Other Names: Clotinab + Thrombuster II
  Arms: Both use

SUMMARY:
The routine use of glycoprotein (Gp) IIb-IIIa inhibitor such as abciximab is not recommended by current ACC/AHA guideline (Class IIb, level of evidence of A). This may be partly due to potential increase of bleeding. Compared bolus injection followed by continuous infusion of Gp IIb-IIIa inhibitor, single bolus administration was proposed to decrease bleeding complication while maintaining decrease ischemic events. It was also reported that direct intracoronary injection of abciximab might be superior to intravenous injection regarding myocardial perfusion.

Aspiration thrombectomy is regarded as important adjunctive therapy in the treatment of acute ST-elevation myocardial infarction (IIa, level of evidence of B). We hypothesized that combination of intracoronary abciximab bolus injection and aspiration thrombectomy might enhance adequate myocardial perfusion in patient with acute ST-elevation myocardial infarction. We will determine whether combination of intracoronary abciximab injection and aspiration thrombectomy is superior to each treatment only in terms of myocardial perfusion through index of microcirculatory resistance and cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between at least 18 years of age and less than 80 years of age.
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving intracoronary abciximab and/or aspiration thrombectomy.
* He/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have evidence of acute ST-segment elevation myocardial infarction with TIMI 0 or 1 flow, or visible thrombi (thrombus grade ≥ 3)
* Target lesion(s) must be located in a native coronary artery in the proximal to mid segment with estimated reference diameter of ≥ 2.5 mm and ≤ 4.0 mm.
* Target lesion(s) must be amenable for percutaneous coronary intervention.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Abciximab, Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.)
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or refuses blood transfusions.
* Baseline hemogram with Hb<10g/dL or PLT count <100,000/μL
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* Patients with severe LV systolic dysfunction (LVEF<25%) or in cardiogenic shock
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Index of microcirculatory resistance by fractional flow reserve (FFR) | 1 day
  Immediate measurement of Index of microcirculatory resistance
Microvascular obstruction by cardiac magnetic resonance | 7 days
  Microvascular obstruction by cardiac magnetic resonance

SECONDARY OUTCOMES:
Final TIMI flow grades | 1 day
  immediate measurement after successful PCI
Final TMP grades | 1 day
  immediate measurement of Final TMP grades
ST-segment resolution on ECG | 1 day
  ST-segment resolution on ECG 90-minute after PCI
Peak troponin I level | 5 days
  Peak troponin I level during hospitalization
target vessel failure | 1 month
  1-month target vessel failure defined as a composite of death from cardiac causes, any MI (not clearly attributable to a non-target vessel), or clinically indicated target vessel revascularization (TLR)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Gyun Ahn, M.D., Principal Investigator — Yonsei University
Locations (1):
- Yonsei University Wonju College of Medicine, Wonju Christian Hospital, Wŏnju, South Korea

REFERENCES:
- [Derived] Ahn SG, Lee SH, Lee JH, Lee JW, Youn YJ, Ahn MS, Kim JY, Yoo BS, Yoon J, Choe KH, Tahk SJ. Efficacy of combination treatment with intracoronary abciximab and aspiration thrombectomy on myocardial perfusion in patients with ST-segment elevation myocardial infarction undergoing primary coronary stenting. Yonsei Med J. 2014 May;55(3):606-16. doi: 10.3349/ymj.2014.55.3.606. Epub 2014 Apr 1. PMID 24719126